CLINICAL TRIAL: NCT03212768
Title: Outcome of Low Energy Ankle Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: LEFA
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Trans-syndesmotic fixation — antromedial approach for medial malleolus fractures, posterolateral or direct lateral approach for fibula fractures, direct fixation of third malleolus by posterior approach, Trans-syndesmotic fixation ,cement augmentation and Tibiotalocalcaneal fusion

SUMMARY:
Ankle fractures are among the most common osseous injuries to the lower extremity, and remain a significant source of morbidity for both the young and the elderly. Recent cross-national studies have shown a significant increase in the incidence and severity of ankle fractures among the elderly population.

ELIGIBILITY:
Inclusion Criteria:

- all types of trumatic ankle fractures due to low energy amenable to surgical open reduction and internal fixation .

Exclusion Criteria:

* previous surgery.
* Disorders of bone metabolism other than osteoprosis (ie, Paget disease , renal osteodystrophy , osteomalacia )
* Patient with moderate or severe congnitive impairment or patients with Parkinson disease or dementia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with Grossly displaced fracture-dislocations
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The rate of recovery from the surgery of fractures | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt